CLINICAL TRIAL: NCT00791349
Title: A Placebo- and Positive-controlled, Randomized Study Evaluating QT and QTc Intervals Following Administration of Immediate-release Paliperidone in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study of QT and QTc Intervals in Patients Administered Immediate Release Paliperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004201
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Mood Disorders; Antipsychotic drugs; Cardiovascular; Immediate release (IR) Paliperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Immediate release (IR) Paliperidone

SUMMARY:
The purpose of this study is to assess the cardiovascular safety of paliperidone in patients with schizophrenia or schizoaffective disorder, with particular attention to the length of the QT/QTc interval, to measure and review other electrocardiogram (ECG) parameters, such as QRS and PR intervals, to explore the relationship between the pharmacokinetics of paliperidone and ECG parameters of interest, and to explore the safety and tolerability of paliperidone

DETAILED DESCRIPTION:
This is a multicenter, placebo- and positive-controlled, randomized study consisting of 3 periods: a screening period of up to 14 days (including a 5-day washout period), a double-blind period of 10 days (including the treatment phase [Days 1 to 8] and the posttreatment phase [Days 9 and 10]), and an end-of-study evaluation. Eligible patients will be randomly assigned to treatment with either paliperidone or moxifloxacin. Patients randomly assigned to receive paliperidone will receive placebo on Day 1, paliperidone 4 mg on Day 2, paliperidone 6 mg on Day 3, and paliperidone 8 mg on Days 4 through 8. Patients assigned to receive moxifloxacin will receive placebo on Days 1 through 7 and moxifloxacin 400 mg on Day 8. The moxifloxacin treatment group will provide a concurrent active control to confirm that the study is adequate to detect a drug effect (i.e., assay sensitivity) on QTc interval. Baseline ECGs will be recorded on the last day of the washout period (Day 1). Serial time matched 12 lead ECG triplicate readings will be recorded on Days 1, 2, 3, 4, 5 (predose), 8, 9, and 10. This study is being conducted to thoroughly assess potential QT/QTc interval changes following administration of paliperidone. The results from this safety study, along with the ECG results from all paliperidone clinical studies, will be used in the evaluation of the cardiovascular safety of paliperidone. Paliperidone IR orally once daily: 4 mg on Day 2, 6 mg on Day 3, and 8 mg on Days 4 through 8; Active control: a single oral dose of moxifloxacin 400 mg on Day 8

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of schizophrenia or schizoaffective disorder as defined by DSM-IV criteria, with no exacerbation of psychosis for at least 3 months prior to screening
* Patients must have a normal 12-lead ECG at screening and on Day -1, including: Normal sinus rhythm (heart rate between 50 and 100 beats per minute)
* QTcB interval < = 430 msec for men, < = 450 msec for women
* QRS interval <110 msec, PR interval < 200 msec
* Patients must weigh > = 50 kg ( > = 110 lb), with a body mass index > = 18 and < = 35 kg/m2
* Female patients must be postmenopausal (for at least 1 year), surgically sterile, or practicing an effective non-hormonal method of birth control (e.g., intrauterine device, double-barrier method, male partner sterilization, abstinence) before entry and throughout the study
* must have a negative serum beta human chorionic gonadotropin pregnancy test at screening
* and must have a negative urine pregnancy test within 24 hours before Day 1 of the randomization period.

Exclusion Criteria:

* Patient meets DSM-IV criteria for psychoactive substance dependence in the 3 months prior to screening
* Patient is at risk for suicidal or violent behavior, as judged by the investigator: Patient has a clinically significant abnormality on ECG at screening or on Day -1 of the study
* Patient has a heart rhythm disturbance that is known or suggested by history or that is demonstrated on ECG at screening
* Patient has a blood pressure outside of the normal range (supine systolic blood pressure <90 or >140 mmHg and/or diastolic blood pressure <60 or > 90 mmHg)
* Patient has unusual T-wave morphology in a majority of leads of the ECG (such as bifid T waves, low T waves) or prominent U waves at screening: Patient has a history of additional risk factors for torsade de pointes, such as heart failure, hypokalemia, family history of known long QT interval syndrome, or sudden unexplained death at a young age ( < = 40 years) in a first-degree relative (i.e., biological parent, sibling, or offspring)
* Patient has a relevant history of any significant and/or unstable cardiovascular, respiratory (including bronchial asthma), neurologic (including seizures or significant cerebrovascular disease), renal, hepatic, endocrine, immunologic, ophthalmologic, hematological, or other systemic disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2005-02; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To assess the cardiovascular safety of paliperidone in schizophrenic or schizoaffective patients, with particular attention to the length of the QT/QTc interval. Other ECG parameters, such as QRS and PR intervals, will also be carefully measured

SECONDARY OUTCOMES:
To explore the relationship between the pharmacokinetics of paliperidone and ECG parameters of interest, and to explore the safety and tolerability of paliperidone

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of QT and QTc intervals in patients administered immediate release paliperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=565&filename=CR004201_CSR.pdf